CLINICAL TRIAL: NCT02717715
Title: The Effect of a Tele-supervised Home Based Rehabilitation Program on Physical Fitness, Quality of Gait, Upper Limb Disability and Quality of Life in People After Chronic Stroke in a Urban Setting in Suriname. Randomised Controlled Trial.
Brief Title: SunRISe Study - Stroke Rehabilitation In Suriname
Acronym: SunRISe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Anton De Kom University (Unknown); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Roselien Buys, Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VG 023-15
Record Dates: First submitted 2016-03-05; First posted 2016-03-24 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Stroke patients from the intervention group will be, on top of usual care, offered a holistic home based and semi-supervised stroke rehabilitation program followed by a period of tele-supervision.
  Interventions: Behavioral: Home base stroke rehabilitation
- Control group (No Intervention): The participants in the control group will only receive usual care.

INTERVENTIONS:
Behavioral: Home base stroke rehabilitation — The intervention consists of physiotherapy exercises targeting functional and physical capacity.
  Arms: Intervention group

SUMMARY:
This study aims to determine the effect of a supervised home-based physical fitness program on the aerobic capacity, quality of gait and health related quality of life in people with chronic ischemic stroke. Secondly, feasibility of the program for implementing a long term lifestyle change will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* ability to understand measurement procedures defined as MMSE >24
* last stroke >6 months ago
* mild to moderate stroke deficit defined by Fugl Meyer test score of 27 to 90 for upper and lower extremities
* FAC ≥3
* medical clearance to participate in a moderate exercise program
* living at home and having a minimum of 5 stairs at home

Exclusion Criteria:

* serious cardiac condition
* other serious end organ damage
* other neurological deficits leading to disability
* uncontrolled blood pressure (systolic pressure >140, diastolic pressure >90)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake | 4 weeks, 8 weeks and 5 months after start of rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Anton De Kom University, Paramaribo, Suriname

IPD SHARING:
Plan to Share IPD: No